CLINICAL TRIAL: NCT06348004
Title: A Study on the Risk of Rebleeding Within 30 Days After Discharge in Patients With Cirrhosis and Acute Variceal Bleeding Following Short-term Albumin Infusion
Brief Title: The Association Between Albumin Administration and Short-term Rebleeding Risk in Cirrhosis Patients With Acute Variceal Hemorrhage and Stable Hemodynamics
Status: Active, not recruiting | Type: Observational
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Han Ma, Dr., Zhejiang University
Other Study IDs: 2024IIT-0125
Record Dates: First submitted 2024-03-28; First posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Cirrhosis; Acute Variceal Haemorrhage
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- albumin user group and albumin non-user group

SUMMARY:
The impact of albumin administration in cirrhotics with acute variceal hemorrhage (AVH) is controversial. We aim to investigate the short-term rebleeding risk associated with albumin administration in a retrospective study of hospitalized cirrhotics with AVH with stable hemodynamics. This retrospective analysis includes clinical data of cirrhosis patients with acute variceal bleeding admitted to our hospital from January 2021 to October 2023. Propensity score matching will be performed to account for potential confounders associated with albumin use for outcome analysis. According to the outcome, patients will be divided into rebleeding group and non-rebleeding group. To investigate the impact of albumin infusion on the rebleeding risk in the propensity-matched cohort, patients will be divided into albumin user group and albumin non-user group. The primary outcome is the rebleeding risk within 30 days after discharge.

ELIGIBILITY:
Inclusion criteria (1) Patients were diagnosed with liver cirrhosis with esophageal and gastric varices; (2) Patients were presented with any evidence or signs of acute upper gastrointestinal bleeding within 3 days before admission, including hematemesis, melena, and positive fecal occult blood. (3) Endoscopy or imaging data suggested the presence of AVB.

Exclusion criteria

(1) Patients with unstable hemodynamics (patients whose sBP<90mmHg or heart rate >120 bpm at admission). (2) Patients who were initially treated at other facilities but later transferred to our hospital without comprehensive medication records. (3) Ages <18 years old or ages >85 years old. (4) Patients with incomplete data.

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Cirrhosis patients with acute variceal bleeding who were admitted to the First Affiliated Hospital, Zhejiang University School of Medicine from January 2021 to October 2023.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
The rebleeding risk within 30 days after discharge. | From enrollment to 30 days after discharge

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China